CLINICAL TRIAL: NCT05590676
Title: A Phase I Safety and Feasibility of Metformin Treatment in Infants After Perinatal Brain Injury
Brief Title: Metformin Treatment in Infants After Perinatal Brain Injury
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Waterloo (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Brian Kalish, Staff Neonatologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3987
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Hypoxic Ischemic Encephalopathy of Newborn; Premature Birth
Keywords: Hypoxic Ischemic Encephalopathy; Newborn; Metformin; Prematurity
MeSH Terms: conditions — Premature Birth; Hypoxia-Ischemia, Brain | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HIE: 20 mg/kg (Experimental)
  Interventions: Drug: Metformin Hydrochloride
- HIE: 25 mg/kg (Experimental)
  Interventions: Drug: Metformin Hydrochloride
- Preterm: 15 mg/kg (Experimental)
  Interventions: Drug: Metformin Hydrochloride
- Preterm: 20 mg/kg (Experimental)
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Infants will receive 14 consecutive doses, once daily, of metformin, with two dose cohorts.
  Arm 1: Five infants with HIE will be enrolled on the first dose cohort of 20 mg/kg. Once complete, another five infants will be enrolled on the second dose cohort of 25 mg/kg.
  Arm 2: Five preterm infants will be enrolled on the first dose cohort of 15 mg/kg. Once complete, another five preterm infants will be enrolled on the second dose cohort of 20 mg/kg.

SUMMARY:
A phase I study to test the feasibility and safety of treatment with metformin in infants affected by hypoxic ischemic encephalopathy (HIE) or prematurity-related brain injury

ELIGIBILITY:
Inclusion Criteria:

HIE Patients:

1. > 35 weeks gestation at time of birth
2. ≤3 months at time of consent
3. Clinical diagnosis of HIE
4. Infant received therapeutic hypothermia for the treatment of HIE
5. Family lives within one hour distance of the Hospital for Sick Children (in order to facilitate home visits)

Preterm Infants:

1. <32 weeks gestation at time of birth
2. 36-44 weeks corrected (postmenstrual) gestational age at time of metformin administration
3. Clinical team anticipates hospitalization at SickKids for at least 1 week after study enrollment

Exclusion Criteria:

1. Have a known genetic or chromosomal disorder.
2. Congenital or acquired liver or kidney disease that might, in the opinion of the Principal Investigator or delegate, affect drug metabolism.
3. History of hypoglycemia in the newborn period requiring glucose infusion rate > 10 mg/kg/min or treatment with glucagon or diazoxide.
4. Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate, interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk
5. >3 months of age at the time of enrollment (term HIE patients only)
6. Weight <10%ile based on WHO growth charts at time of initiation of study drug (term HIE patients only).
7. Maternal use of metformin while actively breastfeeding.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with hypoglycemia (serum glucose <3.3mmol/L) | 2 weeks
  Number of patients with hyperglycemia (glucose>10mmol/L)

SECONDARY OUTCOMES:
Plasma metformin levels | 2 weeks
  Pharmacokinetics analysis
Number of patients who complete study | 2 weeks
  Feasibility of study intervention administration
Number of patients who complete all study procedures | 2 weeks
  Feasibility of executing study operations

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Kalish, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontartio, Canada